CLINICAL TRIAL: NCT05053646
Title: Biological Augmentation Of Meniscal Repair With Marrow Venting: A Randomized Controlled Trial
Brief Title: This is a Study to Verify if Marrow Venting Procedure Can Improve Meniscal Suture Healing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Candrian (Other)
Responsible Party: Sponsor-Investigator, Christian Candrian, Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORL-ORT-019
Record Dates: First submitted 2021-07-22; First posted 2021-09-22 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Meniscal Tear

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Marrow venting arm (Experimental): Meniscal suture associated with marrow venting procedure
  Interventions: Procedure: Meniscal repair; Procedure: Marrow venting procedure
- Control arm (Active Comparator): Meniscal suture alone, without marrow venting procedure
  Interventions: Procedure: Meniscal repair

INTERVENTIONS:
Procedure: Meniscal repair — The meniscus is trimmed with an arthroscopic punch followed by an electric shaver to expose the margins of the tear and remove damaged tissue. Vertical sutures are made using TRUESPAN™ Meniscal Repair System (DePuy Synthes) to approximate both the femoral and tibial surfaces of the torn meniscus.
Procedure: Marrow venting procedure — After meniscal repair, a bone marrow venting procedure will be performed: a 45° micro-fracture awl is repeatedly penetrated through the bone of the intercondylar notch at the PCL origin until marrow elements are seen to enter the joint.
  Arms: Marrow venting arm

SUMMARY:
Meniscal suture represents the current surgical practice, and marrow venting is a low risk procedure. Bone venting may be able to improve the outcome of meniscal repair, allowing the patient a better recovery.

DETAILED DESCRIPTION:
Meniscal tears are one of the most common lesions of the knee and are a risk factor for the development of knee osteoarthritis. A meniscal tear commonly causes knee pain, stiffness, loss of function and sometimes catching or locking of the knee, affecting patients' ability to participate in their everyday activities. In case of ineffective conservative management, meniscal tears are treated with meniscectomy (partial or total) or meniscal repair, with the latter considered, when possible, the optimal choice.

Meniscal repair consists of a suture that juxtaposes the flaps of the injured meniscus to facilitate the healing of the tear. Unfortunately, meniscal healing capability is limited. A higher rate of meniscal tears healing has been documented in patients treated simultaneously with a meniscal repair and anterior cruciate ligament reconstruction. A surgical augmentation technique performing micro-fractures on the medial aspect of the lateral femoral condyle during meniscal repair surgery has been developed to mimic the beneficial effect of anterior cruciate ligament reconstruction on the joint environment. This technique has been successfully tested in preclinical studies, in human cohort studies and, recently, in a randomized control trial. However, these randomised controlled trials present some methodological weaknesses, such as a low number of included patients, and included only full-thickness vertical longitudinal tears in the red-red zone, the meniscal tears with the highest healing potential. The effect of additional micro-fractures on the healing capacity of meniscal tears involving the red-white zone has never been tested.

ELIGIBILITY:
Inclusion Criteria:

* Arthroscopic confirmed suturable meniscal tears,
* Monolateral meniscal tears,
* 18-45 years,
* BMI>18,5 and <35 kg/m2,
* Ability to give informed consent by signature.

Exclusion Criteria:

* Bilateral meniscal tears requiring treatment,
* Associated ligament lesions requiring treatment,
* Associated cartilage lesions (Outerbridge > 2),
* Knee axis deformities requiring correction
* Generalized ligamentous laxity,
* Radiographic knee ostheoarthritis,
* Other reasons for knee pain,
* Pregnant or lactating women,
* Serious systemic diseases such as cardiac, hepatic or renal failure, rheumatic diseases, non-compensated diabetic, psychological illnesses, central or peripheral neurological diseases, and autoimmune diseases,
* Enrolled in another ongoing clinical trial.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-29 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
subjective International Knee Documentation Committee (IKDC) score | 2 years
  evaluated subjective IKDC score 2-years after intervention in two groups

SECONDARY OUTCOMES:
Objective International Knee Documentation Committee (IKDC) | (pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years)
  Objective IKDC - International Knee Documentation Committee (pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years)
Lysholm score (pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years) | (pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years)
  Lysholm score (pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years)
Knee Injury and Osteoarthritis Outcome Score - KOOS | (pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years)
  Knee Injury and Osteoarthritis Outcome Score - KOOS (pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years)
Pain 0-10 Numerical Rating Scale (NRS) | (pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years)
  Pain 0-10 numerical rating scale - NRS (pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years)
Function 0-10 Numerical Rating Scale (NRS) | (pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years)
  Function 0-10 numerical rating scale - NRS (pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years)
Tegner score | (prior to the injury (e.g. referred to the day before), pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years)
  Tegner score (prior to the injury (e.g. referred to the day before), pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years)
Healing rate | 1 year
  Healing rate (MRI at 1 year)
Treatment related adverse events | 5 years
  Treatment related adverse events: overall, intra-operative, short- (<3 months), mid- (3 months, 2 years), long-term (>2 years) adverse events
Function curves during the first 6 weeks. | 6 weeks
  Function curves during the first 6 weeks.
Pain curves during the first 6 weeks. | 6 weeks
  Pain curves during the first 6 weeks as retrieved by the values produced with the EOC EMApp.
Radiographic progression of knee osteoarthritis | 5 years
  Radiographic progression of knee osteoarthritis (x-ray at 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Candrian, MD, Principal Investigator — Ente Ospedaliero Cantonale, Bellinzona
Locations (2):
- Switzerland (2):
  - Ente Ospedaliero Cantonale, Lugano
  - Clinica Ars Medica, Lugano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn JH, Kwon OJ, Nam TS. Arthroscopic repair of horizontal meniscal cleavage tears with marrow-stimulating technique. Arthroscopy. 2015 Jan;31(1):92-8. doi: 10.1016/j.arthro.2014.07.029. Epub 2014 Sep 18. PMID 25242513
- [Background] Briggs KK, Kocher MS, Rodkey WG, Steadman JR. Reliability, validity, and responsiveness of the Lysholm knee score and Tegner activity scale for patients with meniscal injury of the knee. J Bone Joint Surg Am. 2006 Apr;88(4):698-705. doi: 10.2106/JBJS.E.00339. PMID 16595458
- [Background] Bryant D, Dill J, Litchfield R, Amendola A, Giffin R, Fowler P, Kirkley A. Effectiveness of bioabsorbable arrows compared with inside-out suturing for vertical, reparable meniscal lesions: a randomized clinical trial. Am J Sports Med. 2007 Jun;35(6):889-96. doi: 10.1177/0363546506298582. Epub 2007 Mar 2. PMID 17337726
- [Background] Charles HC, Kraus VB, Ainslie M, Hellio Le Graverand-Gastineau MP. Optimization of the fixed-flexion knee radiograph. Osteoarthritis Cartilage. 2007 Nov;15(11):1221-4. doi: 10.1016/j.joca.2007.05.012. Epub 2007 Oct 31. PMID 17977754
- [Background] Crawford K, Briggs KK, Rodkey WG, Steadman JR. Reliability, validity, and responsiveness of the IKDC score for meniscus injuries of the knee. Arthroscopy. 2007 Aug;23(8):839-44. doi: 10.1016/j.arthro.2007.02.005. PMID 17681205
- [Background] de Girolamo L, Galliera E, Volpi P, Denti M, Dogliotti G, Quaglia A, Cabitza P, Corsi Romanelli MM, Randelli P. Why menisci show higher healing rate when repaired during ACL reconstruction? Growth factors release can be the explanation. Knee Surg Sports Traumatol Arthrosc. 2015 Jan;23(1):90-6. doi: 10.1007/s00167-013-2712-8. Epub 2013 Oct 22. PMID 24146050
- [Background] Dean CS, Chahla J, Matheny LM, Mitchell JJ, LaPrade RF. Outcomes After Biologically Augmented Isolated Meniscal Repair With Marrow Venting Are Comparable With Those After Meniscal Repair With Concomitant Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2017 May;45(6):1341-1348. doi: 10.1177/0363546516686968. Epub 2017 Feb 1. PMID 28298056
- [Background] Ding C, Martel-Pelletier J, Pelletier JP, Abram F, Raynauld JP, Cicuttini F, Jones G. Meniscal tear as an osteoarthritis risk factor in a largely non-osteoarthritic cohort: a cross-sectional study. J Rheumatol. 2007 Apr;34(4):776-84. Epub 2007 Mar 15. PMID 17361984
- [Background] Driscoll MD, Robin BN, Horie M, Hubert ZT, Sampson HW, Jupiter DC, Tharakan B, Reeve RE. Marrow stimulation improves meniscal healing at early endpoints in a rabbit meniscal injury model. Arthroscopy. 2013 Jan;29(1):113-21. doi: 10.1016/j.arthro.2012.06.023. Epub 2012 Nov 30. PMID 23200846
- [Background] Englund M, Guermazi A, Roemer FW, Aliabadi P, Yang M, Lewis CE, Torner J, Nevitt MC, Sack B, Felson DT. Meniscal tear in knees without surgery and the development of radiographic osteoarthritis among middle-aged and elderly persons: The Multicenter Osteoarthritis Study. Arthritis Rheum. 2009 Mar;60(3):831-9. doi: 10.1002/art.24383. PMID 19248082
- [Background] Englund M, Roemer FW, Hayashi D, Crema MD, Guermazi A. Meniscus pathology, osteoarthritis and the treatment controversy. Nat Rev Rheumatol. 2012 May 22;8(7):412-9. doi: 10.1038/nrrheum.2012.69. PMID 22614907
- [Background] Freedman KB, Nho SJ, Cole BJ. Marrow stimulating technique to augment meniscus repair. Arthroscopy. 2003 Sep;19(7):794-8. doi: 10.1016/s0749-8063(03)00695-9. PMID 12966391
- [Background] Howarth WR, Brochard K, Campbell SE, Grogan BF. Effect of Microfracture on Meniscal Tear Healing in a Goat (Capra hircus) Model. Orthopedics. 2016 Mar-Apr;39(2):105-10. doi: 10.3928/01477447-20160119-04. Epub 2016 Jan 25. PMID 26811956
- [Background] Kaminski R, Kulinski K, Kozar-Kaminska K, Wasko MK, Langner M, Pomianowski S. Repair Augmentation of Unstable, Complete Vertical Meniscal Tears With Bone Marrow Venting Procedure: A Prospective, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study. Arthroscopy. 2019 May;35(5):1500-1508.e1. doi: 10.1016/j.arthro.2018.11.056. Epub 2019 Mar 20. PMID 30902532
- See also: Common Terminology Criteria for Adverse Events (CTCAE) — https://www.eortc.be/services/doc/ctc/CTCAE_4.03_2010-06-14_QuickReference_5x7.pdf
- See also: 7. Ordinance on Clinical Trials in Human Research (ClinO) — http://www.admin.ch/opc/de/classified-compilation/20121176/index.html